CLINICAL TRIAL: NCT05749601
Title: Study of Anatomical and Imaging Characteristics in Relation With the Risk Factors Involved in KOA Progression
Brief Title: Risk Factor Involved in Knee Osteoarthritis (KOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iacob Czihac Emergency Military Clinical Hospital (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10/A575
Record Dates: First submitted 2022-10-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — ETV3 protein, human; Reactive Nitrogen Species

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Patients without knee osteoarthritis (KOA) grade 0 (Active Comparator): Patient without knee affection
  Interventions: Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid; Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis; Other: The influence of ROS from the synovial fluid on the severity of KOA
- Patients with KOA grade I (Experimental): Kellgren-Lawrence classification (KL) grade I- doubtful narrowing of the joint space and possible osteophytes
  Interventions: Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid; Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis; Other: The influence of ROS from the synovial fluid on the severity of KOA
- Patients with KOA grade II (Experimental): KL grade II - definite osteophytes and possible narrowing of joint space.
  Interventions: Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid; Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis; Other: The influence of ROS from the synovial fluid on the severity of KOA
- Patients with KOA grade III (Experimental): KL grade III- definite narrowing of the joint space, significant osteophytosis, and possible bone deformities.
  Interventions: Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid; Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis; Other: The influence of ROS from the synovial fluid on the severity of KOA
- Patients with KOA grade IV (Experimental): KL grade IV- marked joint space narrowing accompanied by deformities, bone sclerosis, and large osteophytes
  Interventions: Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid; Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis; Other: The influence of ROS from the synovial fluid on the severity of KOA

INTERVENTIONS:
Other: Influence of the metabolic syndrome (MetS) parameters on knee osteoarthritis (KOA) severity, the assesment of the reactive oxygen species and reactive nitrogen species in knee synovial fluid — Highlighting the influence of environment of origin on KOA incidence and corelated impact of high-density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol, triglycerides and body mass index (BMI). The analytes from synovial fluid were determined by fluorometric method.
Other: The influence of patellofemoral morphology in the radiological severity of knee osteoarthritis — Highlighting the influence of distal femoral torsion angle, patellofemoral congruence angle and sulcus angle, in KOA severity under the influence of sex and age.
Other: The influence of ROS from the synovial fluid on the severity of KOA — Highlighting the influence of ROS from the synovial fluid in KOA severity under the influence of some biochemicals blood constants.

SUMMARY:
Clinical study regarding the incidence and severity of knee osteoarthritis (KOA) in a certain area from South-Eastern Europe. Aim of the clinical study: to determine the KOA grade through X-Ray studies, to perform nuclear magnetic resonance (NMR) analysis to assess the KOA severity and to determine the level of significant parameters in the synovial liquid extracted from the patients presenting KOA.

DETAILED DESCRIPTION:
Clinical study regarding the incidence and severity of KOA in a certain area from South-Eastern Europe. Clinical study on 85 patients out 373 participants that were screened, chosen based on inclusion/exclusion criteria.

Aim of the clinical study: to determine the KOA grade through X-Ray studies, to perform nuclear magnetic resonance (NRM) analysis to assess the KOA severity. Data corroboration of the KOA degree with the results of the blood samples analysis, looking for the influence of the metabolic syndrome (MetS) parameters - high-density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol, triglycerides, glycemia, and then the body mass index (BMI). In the meantime, there is intended to associate the environment of origin of the patients from the trial group with the KOA incidence and severity. To determine the level of significant parameters in the synovial liquid extracted from the patients presenting KOA, analysis of the degradation products present in the synovial fluid of patients with KOA, such as free radicals, like reactive oxygen species (ROS) and reactive nitrogen species (RNS) and their influence on the severity of the pathology.

ELIGIBILITY:
Inclusion Criteria:

* male and female with knee pain (complaints); presented symptoms and clinical signs corresponding to KOA and had knee X-rays in the anteroposterior view and nuclear magnetic resonance (NMR) performed for setting the diagnosis with unilateral or bilateral knee pain; patients with clinically determined and recorded values of total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides and the glycemia in the clinical observation sheet.

Exclusion Criteria:

* patients presenting lower limb arthroplasties; history of lower limb or pelvis fractures and previous knee surgery: ligamentoplasty, meniscectomy; inflammatory rheumatic diseases such as rheumatoid polyarthritis; other major conditions like malignant illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
The influence of metabolic syndrome parametres and environment of origin in KOA severity | up 2 weeks
  In this part of the study I included 85 patients for whom I measure the parameters of the metabolic syndrome: a high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglyceride, total cholesterol and body mass index (BMI) and I made the corelation of knee osteoarthritis (KOA) Kellgren-Lawrence radiological classification (KL). The formula form BMI was kg/ m2. I raported the influence of the environment of origin in relation to the severity of KOA, performing the statistical analysis of the obtained data, applied metod ANOVA, specific ordinal and binomial logistic regression models, p value <0,005. 95% confidence interval, without non-inferiority/equivalence test.

SECONDARY OUTCOMES:
The influence of patellofemoral morphology in KOA severity | 1 week
  I measured distal femoral torsion angle, patellofemoral congruence angle and sulcus angle for 43 patients who had NRM examinations and I raported their impact in KOA severity under the influence of sex and age.

OTHER OUTCOMES:
The influence of reactive oxygen species (ROS) level in KOA severity | 3 weeks
  In this analysis, 28 patients were included and I studied the average of 3 determinations of ROS from the synovial fluid using the OxiSelectTM kit and their impact in KOA severity under the influence of some biochemicals blood constants.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoleta B Tudorachi, MD, Principal Investigator — "Ovidius" University of Constanța, Romania
Locations (1):
- 3 "Iacob Czihac" Emergency Military Clinical Hospital, 7-9 General Henri Mathias Berthelot St., 700483 Iasi, Romania, Iași, Romania

IPD SHARING:
Plan to Share IPD: No